CLINICAL TRIAL: NCT03884309
Title: Tolerance, Compliance and Growth of Infants Fed an Extensively Hydrolyzed Infant Formula With Added Human Milk Oligosaccharides
Brief Title: Evaluation of Infants Fed an Extensively Hydrolyzed Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL32
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Protein Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Hydrolyzed Protein Infant Formula (Experimental): hydrolyzed protein infant formula powder in cans
  Interventions: Other: Experimental Hydrolyzed Protein Infant Formula

INTERVENTIONS:
Other: Experimental Hydrolyzed Protein Infant Formula — fed ad libitum

SUMMARY:
This is a single group, non-randomized, multicenter study to assess the effects of a hypoallergenic casein hydrolysate powdered infant formula on gastrointestinal (GI) tolerance, growth and compliance in an intended use infant population.

ELIGIBILITY:
Inclusion Criteria:

* Participant is presently consuming an extensively hydrolyzed infant formula (EHF) for persistent feeding intolerance symptoms, symptoms of suspected food protein (milk and/or soy) sensitivity, or other conditions where EHF is deemed an appropriate feeding.
* Parent(s) of infants confirm their intention not to administer prescription medications, over the counter medications, home remedies, prebiotics, probiotics, herbal preparations or rehydration fluids that might affect GI tolerance.
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study.
* Parent(s) confirm their intention not to administer vitamins, minerals (with the exception of Vitamin D supplements), solid foods or juices to their infant from enrollment through the duration of the study.
* Participant's parent(s) or a legally authorized representative (LAR) has voluntarily signed and dated an informed consent form (ICF) approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* An adverse maternal, fetal or participant medical history that is thought by the investigator to have potential for effects on growth, and/or development.
* Participant is receiving oral or inhaled steroids.
* Participant participates in another study that has not been approved as a concomitant study.
* Participant has an allergy or intolerance to any ingredient in the study product.
* Participant has been treated with antibiotics or other medications that in the opinion of the PI may affect growth, GI tolerance and/or development, within 2 weeks prior to enrollment.

Max Age: 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Weight for Age | Study Day 1 to Study Day 60
  Change in weight for age z-score

SECONDARY OUTCOMES:
Gastrointestinal Tolerance | Study Day 1 to Study Day 60
  Parent completed diary questions
Length | Study Day 1 to Study Day 60
  Gain measured in cm
Head Circumference | Study Day 1 to Study Day 60
  Gain measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Marriage, PhD, RD, Study Chair — Abbott Nutrition
Locations (6):
- United States (6):
  - Paramount Research Solutions, College Park, Georgia
  - Michael W. Simon, M.D., PSC, Nicholasville, Kentucky
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Memphis & Shelby County Pediatric Group, Memphis, Tennessee
  - Ventavia Research Group, LLC, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas

IPD SHARING:
Plan to Share IPD: Undecided